CLINICAL TRIAL: NCT02712151
Title: Efficacy of Ultrasound-Guided Transversus Abdominis Plane Block for Postoperative Pain Control in Laparoscopic Cholecystectomy: Prospective Randomized Controlled Trial in Pediatric Patients
Brief Title: Efficacy of Transversus Abdominis Plane Block for Laparoscopic Cholecystectomy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Karen Boretsky, Dr. Karen Boretsky, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-P00022058
Record Dates: First submitted 2016-03-08; First posted 2016-03-18 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative
Keywords: transversus abdominal plane block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal Wall Block with Ropivacaine 0.2% (Active Comparator): Patients will receive bilateral transversus abdominis plane and rectus sheath blocks via ultrasound guidance. A total of 1.0ml/kg distributed between the four blocks (0.4+0.4+0.1+0.1) of 0.2% Ropivacaine (max 50ml) will be injected, as a one time single shot injection, into the fours sites. Surgical infiltration of the four port sites will receive 0.4ml/kg of sterile saline.
  Interventions: Procedure: Abdominal Wall Block; Procedure: Surgical infiltration; Drug: Sterile saline; Drug: Ropivacaine 0.2%; Device: Ultrasound
- Surgical Infiltration with Ropivacaine 0.5% (Active Comparator): Patients will receive surgical infiltration of local anesthetic into the 4 laparoscopic port sites. A total of 0.4 ml/kg (0.1+0.1+0.1+0.1) of 0.5% Ropivacaine, divided between the four port sites (max 20 ml), will be used. A total of 1ml/kg, divided between the TAP (0.4ml/kg on each side) and RS (0.1ml/kg on each side), of sterile saline will be used for the nerve blocks.
  Interventions: Procedure: Abdominal Wall Block; Procedure: Surgical infiltration; Drug: Sterile saline; Device: Ultrasound; Drug: Ropivacaine 0.5%

INTERVENTIONS:
Procedure: Abdominal Wall Block — bilateral TAP and RS blocks.
Procedure: Surgical infiltration — distributed between the 4 laparoscopic port sites.
Drug: Sterile saline — Placebo injection
Drug: Ropivacaine 0.2% — Ropivacaine 0.2% 1.0 ml/kg total in divided doses for bilateral TAP and RS blocks.
  Arms: Abdominal Wall Block with Ropivacaine 0.2%
Device: Ultrasound — For nerve localization
Drug: Ropivacaine 0.5% — Ropivacaine 0.5% 0.4 ml/kg total in divided doses distributed between the 4 laparoscopic port sites
  Arms: Surgical Infiltration with Ropivacaine 0.5%

SUMMARY:
Laparoscopic cholecystectomy is associated with considerable postoperative pain and surgeon-administered local anesthetic infiltration is the standard practice for achieving post-operative analgesia. However, recent studies have shown that pediatric patients continue to experience significant pain during the first 24 hours.

The investigators plan to conduct a prospective, double-blinded, randomized study where patients will be designated into either a test group receiving an ultrasound-guided transversus abdominis plane (TAP) and rectus sheath (RS) blocks with ropivacaine and peri-portal sterile saline or the control group that will receive ultrasound-guided TAP block with sterile saline and peri-portal infiltration of ropivacaine. The anesthesia team and surgical team will both be blinded as well as the research personal in the postoperative period. Patients age 5-17 and American Society of Anesthesiology status I and II undergoing laparoscopic cholecystectomy will be included.

The study hypothesis is that ultrasound-guided peripheral nerve blocks, specifically single shot transversus abdominis plane and rectus sheath blocks, are superior to local wound infiltration during laparoscopic cholecystectomy for decreasing postoperative pain and pain related behavior and facilitating functional recovery.

DETAILED DESCRIPTION:
Patients will be randomized into either a test group receiving an ultrasound-guided TAP block with ropivacaine and peri-portal sterile saline or the control group that will receive ultrasound-guided TAP block with sterile saline and peri-portal infiltration of ropivicaine. All patients, who are scheduled to undergo laparoscopic cholecystectomy who meet the inclusion/exclusion criteria, and their parent(s)/guardian(s) will be called by the study staff the afternoon before surgery, who will follow a study script introducing the project and providing them with an opportunity to enroll in this study or opt out. If the patient cannot be reached the day before surgery, they will be offered the opportunity to enroll the day of surgery in the pre-operative holding area. If the decision is made to participate in the study, a physician study investigator will obtain appropriate consent and assent when applicable. Recruitment materials will be provided, if desired. A copy of this consent form will be placed in the Boston Children's Hospital medical record and a separate research record.

Stratified randomization of patients will be conducted by the pharmacy to maintain the double-blinded nature of the study. The pharmacy staff will deliver a study syringe labeled "regional" and a study syringe labeled "local". Depending on randomization, the "regional" syringe will be filled with either ropivacaine 0.2% or normal saline to the corresponding volume based on the dosing outlined. Similarly, the local syringe will be filled with the opposite solution. Thus, if the "regional" syringe is filled with ropivacaine, the local syringe will be filled with normal saline, and vice versa.

Both surgical and anesthesia teams will be blind to the intervention received by the patient.

The patients will be divided into two groups: 1. Abdominal Wall Block with Ropivacaine and 2. Surgical infiltration with Ropivacaine.

The abdominal wall block group will receive: bilateral transversus abdominis plane and rectus sheath blocks via ultrasound guidance. A total of 1.0ml/kg distributed between the four blocks (0.4+0.4+0.1+0.1) of 0.2% Ropivacaine (max 50ml) will be injected, as a one time single shot injection, into the fours sites. Surgical infiltration of the four port sites will receive 0.4ml/kg of sterile saline.

The surgical infiltration group will receive: surgical infiltration of local anesthetic into the 4 laparoscopic port sites. A total of 0.4 ml/kg (0.1+0.1+0.1+0.1) of 0.5% Ropivacaine, divided between the four port sites (max 20 ml), will be used. A total of 1ml/kg, divided between the TAP (0.4ml/kg on each side) and RS (0.1ml/kg on each side), of sterile saline will be used for the nerve blocks.

Intra-operative Methods: After induction of anesthesia, but before the first incision, each patient will receive an ultrasound-guided block by the regional anesthesiologist as follows:

A. Block Placement:

a. Time out performed for procedure b. Site prepared using aseptic technique c. Localization of the bilateral posterior TAP plane and bilateral rectus sheaths using a portable ultrasound machine i. Aseptic preparation of probe with sterile sheath ii. 38mm linear probe (BK Medical, USA) iii. 15 MegaHertz frequency d. Needle: 22g 80mm echogenic e. Drug administration per protocol and group allocation

B. Periportal Infiltration:

a. Injection of drug and volume per protocol into the planned insertion sites for the 4 ports.

All patients will receive acetaminophen IV 15 mg/kg, dexamethasone 0.1 mg/kg, and morphine 0.05 mg/kg after induction of anesthesia but prior to the first incision. At the conclusion of surgery, prior to emergence, each patient will receive ketorolac IV 0.5 mg/kg (max 30 mg). All intraoperative details of care including vitals signs, medication administration, complications, and timing of events are recorded in the electronic anesthesia record.

PACU Methods: Pain will be assessed post-operatively in the PACU (Post-Anesthesia Care Unit) using the FLACC, FACES Pain Rating Scale or Numeric Rating Scale (NRS) as per PACU protocol and as appropriate to patient age. Once the patient is awake and able to respond to questions, a pain score will be obtained and documented by a study investigator until discharge from the recovery room. Morphine 0.05 mg/kg IV will be administered for NRS, FLACC, or FACES score greater than 4. This can be repeated every 10 minutes to a total of 4 doses. Doses, times, and types of all medications administered in the PACU, in addition to the duration of time a patient spends in the PACU, are documented in the electronic medical record (per standard PACU protocol). Post-anesthetic complications are documented by the PACU nurse in the electronic medical record. Trained research personnel will evaluate for the presence or absence of periumbilical analgesia prior to discharge from PACU. The patient will be discharged from the PACU to an in-patient bed when standard PACU discharge criteria are met.

Inpatient Methods: All patients will receive standard postoperative orders to include acetaminophen 15 mg/kg IV q 6 hours, ketorolac 0.5 mg/kg IV q6 hours, morphine 0.05 mg/kg IV q 2 hours as needed, and oxycodone 0.15 mg/kg PO Q 4 hours as needed. Pain will be assessed by the unit nurses using the appropriate scale for age. Morphine 0.5 mg/kg IV or oxycodone 0.15mg/kg will be administered for NRS, FLACC, or FACES score greater than 4.

Pain Scores will be recorded at 3,6,12 and 24 hours postoperatively with the patient at rest and during coughing.

On the morning of POD #1, trained research personnel will administer the appropriate survey of functional recovery. Validated questionnaires to assess postoperative recovery are available for use in pediatric patients < 12 yrs age (Parents Postoperative Pain Management (PPPM)) and adult patients (Post Discharge Surgical Recovery (PDSR) scale (10-13)). No validated survey exists for patients between the ages of 12 -17 and it was decided to extend the PPPM for use on patients up to and including patients 15 years of age and to use the PDSR on any patient older than 15.

In addition, parents and patients will fill out a bedside diary in the form of a bingo card (addendum 2).

Total intravenous and oral opioid (oral oxycodone or other oral opioid given will be converted to IV morphine equivalents).

Doses, times, and types of all medications administered while in the OR, PACU and inpatient units will be abstracted from the patient's electronic medical record soon after the patient is discharged from the hospital to ensure that study protocols were followed. Fentanyl administration will be analyzed separate from other opioids due to its comparatively divergent half-life and potency. Other data related to hospital stay such as length of procedure (surgery start time to surgery stop time), length of time in the OR, length of time in the recovery room, and length of hospital stay, will be also be collected. Any complication or opioid-related side effect will also be collected. Data will be kept in an excel spreadsheet. The spreadsheet will have anonymous patient identifiers and will be kept in a folder on a password protected hard-drive. Only persons involved in the research study will have access to the folder.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 5-17 years old at time of surgery
2. ASA status 1-2
3. Parent is able to provide informed consent and patient's > age 7 able to give assent
4. Patients scheduled for laparoscopic cholecystectomy
5. Surgery will involve and be limited to laparoscopic cholecystectomy
6. Admission status: 24-hour admission to hospital

Exclusion Criteria:

1. Non-English speaking parents/patient.
2. All emergency laparoscopic cholecystectomies or conversion to an open procedure
3. Patients who will remain intubated or require ICU care postoperatively
4. Significant liver or renal disease
5. Coagulopathy
6. Underlying neurocognitive disorder or developmental delay affecting ability to convey feelings of pain to medical staff
7. Diagnosis of chronic pain syndrome
8. Active infection over nerve block sites
9. History of allergy to local anesthetic agents or non-steroidal anti-inflammatory drugs (NSAIDS)
10. Known alcohol or substance abuse within the past 6 months
11. Daily Opioid use
12. ASA class 3 or higher

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
cumulative opioid consumption (both intravenous and enteral) during the perioperative period | 24 hours

SECONDARY OUTCOMES:
post-operative patient-reported pain scores upon arrival to the post-operative care unit and inpatient unit | every eight hours thereafter on the hospital floor for total of 24 hours postoperatively
post-operative episodes of opioid-related side effects, such as nausea, vomiting, constipation, urinary retention, and pruritis | 24 hours
time to first liquid and/or solid PO intake | 24 hours
time to mobilization out of bed | 24 hours
overall patient functional recovery evidenced by validated patient surveys | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karen Boretsky, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finley AG, McGrath PJ, Forward PS, McNeill G, Fitzgerald P. Parents' management of children's pain following 'minor' surgery. Pain. 1996 Jan;64(1):83-87. doi: 10.1016/0304-3959(95)00091-7. PMID 8867249
- [Result] Joshi GP, Beck DE, Emerson RH, Halaszynski TM, Jahr JS, Lipman AG, Nihira MA, Sheth KR, Simpson MH, Sinatra RS. Defining new directions for more effective management of surgical pain in the United States: highlights of the inaugural Surgical Pain Congress. Am Surg. 2014 Mar;80(3):219-28. PMID 24666860
- [Result] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Result] Joshi GP, Kehlet H. Procedure-specific pain management: the road to improve postsurgical pain management? Anesthesiology. 2013 Apr;118(4):780-2. doi: 10.1097/ALN.0b013e31828866e1. No abstract available. PMID 23388191
- [Result] Kluivers KB, Riphagen I, Vierhout ME, Brolmann HA, de Vet HC. Systematic review on recovery specific quality-of-life instruments. Surgery. 2008 Feb;143(2):206-15. doi: 10.1016/j.surg.2007.08.017. Epub 2007 Dec 21. PMID 18242337
- [Result] Kleinbeck SV. Self-reported at-home postoperative recovery. Res Nurs Health. 2000 Dec;23(6):461-72. doi: 10.1002/1098-240X(200012)23:63.0.CO;2-S. PMID 11130605
- [Result] Chambers CT, Reid GJ, McGrath PJ, Finley GA. Development and preliminary validation of a postoperative pain measure for parents. Pain. 1996 Dec;68(2-3):307-13. doi: 10.1016/s0304-3959(96)03209-5. PMID 9121819
- [Result] von Baeyer CL, Chambers CT, Eakins DM. Development of a 10-item short form of the parents' postoperative pain measure: the PPPM-SF. J Pain. 2011 Mar;12(3):401-6. doi: 10.1016/j.jpain.2010.10.002. Epub 2010 Dec 17. PMID 21167790